CLINICAL TRIAL: NCT07282197
Title: Efficacy and Safety Evaluation of Darolutamide+ADT Adjuvant After Radical Prostatectomy (RP) Without ePLND, in High-risk Prostate Cancer Patients Based on Briganti 2019 Nomogram: A Phase II, Single-center, Single-arm, Prospective Study
Brief Title: Darolutamide+ADT Post-RP w/o ePLND in hrPC: Briganti 2019
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23096
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daro+ADT (Experimental): High-risk prostate cancer patients (Briganti 2019 monogram criteria) who did not undergo extended pelvic lymph node dissection (ePLND), will receive Darolutamide 600 mg bid + ADT for 12 months within 12 weeks after RP.
  Interventions: Drug: Darolutamide (BAY 1841788)

INTERVENTIONS:
Drug: Darolutamide (BAY 1841788) — Darolutamide 600 mg bid + ADT x 12 months

SUMMARY:
The goal of this clinical trial is to evaluate whether adjuvant darolutamide plus androgen-deprivation therapy (ADT) can reduce post-operative recurrence and improve disease control in high-risk prostate cancer patients-defined by the Briganti 2019 nomogram-who have undergone radical prostatectomy (RP) without extended pelvic lymph node dissection (ePLND). The main questions it aims to answer are:

1. What proportion of participants remains biochemical-recurrence-free at 2 years, using NCCN criteria (PSA increase >0.1 ng/mL above post-treatment nadir confirmed by two tests ≥2 weeks apart)?
2. What proportion of participants is the 2-year radiographic progression-free survival (rPFS)?

Additional key outcomes include:

* PSA undetectable rates at 6, 12, and 24 months (PSA <0.01 ng/mL).
* Safety and tolerability assessed by CTCAE v5.0.
* Exploratory** patient-reported outcomes: urinary symptoms (IPSS) and quality of life (EQ-5D-3L).

Study type & design: Phase II, single-center, single-arm, prospective interventional study. Enrollment occurs within 12 weeks after RP. ADT is delivered with a GnRH agonist (physician's choice); orchiectomy is excluded. Target sample size is approximately 40 participants; the statistical plan uses a one-sample log-rank framework. Primary and secondary endpoints are assessed over 2 years.

Participants will: Provide informed consent and undergo eligibility confirmation (high-risk per Briganti 2019; post-RP without ePLND; enrollment ≤12 weeks after surgery). Receive darolutamide + ADT according to protocol (GnRH agonist; no orchiectomy). Attend scheduled visits for PSA monitoring, safety labs, and adverse-event assessments (CTCAE v5.0). Undergo radiologic evaluations as per protocol to determine rPFS (RECIST 1.1/PCWG3). Complete IPSS and EQ-5D-3L questionnaires at specified time points to assess urinary symptoms and quality of life.

Primary endpoint: 2-year biochemical-recurrence-free rate. Key secondary endpoints: 2-year rPFS; PSA <0.01 ng/mL at 6/12/24 months; treatment-emergent adverse events.

Exploratory endpoints: IPSS and EQ-5D-3L changes over 2 years.

This trial aims to balance oncologic control with quality of life in a population for whom the therapeutic value of ePLND remains uncertain, by testing whether early adjuvant darolutamide + ADT after RP can meaningfully delay recurrence and progression while maintaining acceptable tolerability.

ELIGIBILITY:
Inclusion Criteria:

* The patient volunteers to participate and signs the informed consent form (ICF);
* Age 18-75 years (inclusive), male;
* Histologically or cytologically confirmed prostatic adenocarcinoma;
* No non-regional lymph-node metastasis, bone metastasis, or other distant metastasis (e.g., visceral) by conventional imaging (bone scan, CT or MRI) or by PET/CT; i.e., M0;
* High-risk per the Briganti 2019 nomogram, i.e., risk >7%;
* PSA <0.1 ng/mL at 6 weeks after radical prostatectomy (RP);
* Has undergone RP without pelvic lymph-node dissection;
* Not suitable for adjuvant/salvage radiotherapy (RT) after RP, or the patient declines RT;
* Patients with lymph-node involvement (LNI) indicated by PSMA-PET who did not undergo extended pelvic lymph-node dissection (ePLND) may be enrolled;
* Patients with negative intraoperative obturator lymph-node biopsy who did not undergo ePLND may be enrolled;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1;
* Adequate hematologic and organ function:

  * Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L (1500/µL);
  * Hemoglobin ≥90 g/L (9.0 g/dL);
  * Platelet count ≥100 × 10⁹/L (100,000/µL) (without transfusion and/or growth factors within 3 months prior to starting study treatment);
  * Serum potassium ≥3.5 mmol/L;
  * Total bilirubin (TBIL) ≤2.0 × ULN (for Gilbert syndrome, TBIL >1.5 × ULN is not eligible; if indirect bilirubin ≤1.5 × ULN, enrollment is allowed);
  * AST and ALT ≤2.5 × ULN;
  * Serum albumin ≥30 g/L (3.0 g/dL);
  * Serum creatinine <2 × ULN;
* Patients of childbearing potential must agree to use effective contraception throughout the study and for 3 months after the last dose.

Exclusion Criteria:

* Histologic features of neuroendocrine differentiation or small-cell carcinoma;
* Prior prostate cancer treatments including any of the following:

  * Systemic therapy, including but not limited to: >2 months of ADT; >2 months of conventional hormonal therapy (e.g., flutamide, bicalutamide); next-generation hormonal agents (e.g., darolutamide, abiraterone, apalutamide, enzalutamide, relugolix); chemotherapy (e.g., docetaxel); immunotherapy; targeted therapy;
  * Local radiotherapy;
* Planned bilateral orchiectomy during the study treatment period;
* Inability to tolerate darolutamide or ADT;
* Concurrent participation in, or planned participation in, another clinical trial;
* A malignancy other than prostate cancer within the past 5 years or concurrently, except for cured basal cell carcinoma of the skin;
* Any concomitant disease or condition that, in the investigator's judgment, presents a serious risk to patient safety, may confound study results, or may interfere with completion of the study (e.g., severe cardiovascular disease, active infection, gastrointestinal disease, neurologic or psychiatric disorders, etc.);
* Any other condition deemed by the investigator to make the patient unsuitable for this study.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who remained biochemical recurrence free for 2 years | 2 years
  biochemical recurrence defined as a PSA increase >0.1 ng/ml above the post-treatment nadir (confirmed by two consecutive measures at least 2 weeks apart), according to NCCN criteria

SECONDARY OUTCOMES:
2-year rate of radiological progression-free survival (rPFS) | 2 years
  rPFS define as the first date of darolutamide+ ADT to the date of first documented radiological progression per RECIST 1.1 for soft tissue or per Prostate Cancer Working Group 3 (PCWG3) for bone lesions, the development of symptoms or complications attributable to cancer progression
6-month/ 12-month/ 24-month PSA undetectable rate | 2 years
  defined as the rate of patients with PSA <0.01 ng/mL
TEAEs | 2 years
  Measured by the number of participants with treatment-related adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0

OTHER OUTCOMES:
Changes in urinary symptoms | 2 years
  International Prostate Symptom Score (IPSS) questionnaire
PRO | 2 years
  EQ-5D-3L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kan Gong, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China